CLINICAL TRIAL: NCT03830658
Title: Effectiveness of a Structured Intervention on the Development of Self-Care Behaviors With Arteriovenous Fistula in Hemodialysis Patients: a Quasi-experimental Study
Brief Title: Effectiveness of a Structured Intervention on the Development of Self-Care Behaviors With AVF in HD Patients
Acronym: SISC-AVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Responsible Party: Principal Investigator, Clemente Neves Sousa, Clinical Professor, Instituto Portugues de Oncologia, Francisco Gentil, Porto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0012
Record Dates: First submitted 2019-01-28; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Arteriovenous Fistula; Hemodialysis
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: The structured intervention designed for this study was a multimethod approach with the purpose of capturing the learning styles of most patients through the use of written, listening and visual learning (10). Structured Intervention on Self-care with AVF (SISC-AVF) has been designed taking into account the structure of care to the person with AVF developed by Sousa (11). The SISC-AVF had the purpose of identifying the signs/symptoms or situations jeopardizing AVF working and includes both a theoretical and a practical part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Intervention on Self-care with AVF (Experimental): The structured intervention designed for this study was a multimethod approach with the purpose of capturing the learning styles of most patients through the use of written, listening and visual learning (10). Structured Intervention on Self-care with AVF (SISC-AVF) has been designed taking into account the structure of care to the person with AVF developed by Sousa (11). The SISC-AVF had the purpose of identifying the signs/symptoms or situations jeopardizing AVF working and includes both a theoretical and a practical part.
  Interventions: Behavioral: Structured Intervention on Self-care with AVF (SISC-AVF)
- Usual-Care Control (Active Comparator): Educational training was given during HD sessions. The dialysis nurse provided information about arteriovenous fistula care and trained the patient when he/she felt it was required. The dialysis units had no documentation concerning the educational training given to patients and the moment to provide such information was not defined, either.
  Interventions: Behavioral: Structured Intervention on Self-care with AVF (SISC-AVF)

INTERVENTIONS:
Behavioral: Structured Intervention on Self-care with AVF (SISC-AVF) — Theoretical Part: structured intervention involved an educational group session with the purpose of teaching patients how to identify situations that can compromise AVF working. Each presentation allowed a maximum of eight patients and took 30 minutes. Each presentation was assessed in the end by asking participants to identify the signs and symptoms of infection, thrombosis and steal syndrome and to describe the care to be taken during dialysis and in the period outside dialysis.
  Practical Part: started a week after the theoretical part, lasting for two weeks, and was given to each participant in an appropriate room at the beginning of the HD treatment. Interactive training sessions were conducted using an informal approach with the objective of developing skills of inspection and palpation of the AVF arm. Inspection had the purpose of enabling participants to identify situations that could compromise the working of the AVF. Each patient was given two 15-minute sessions.

SUMMARY:
End stage renal disease patients (ESRD) should be educated to take care of their arteriovenous fistula (AVF). Educational programs should have clear objectives and the interventions should be well defined. Therefore, assessing the interventions that can have the strongest impact on the patient's acquisition of self-care behaviors with AVF is extremely important. The aim is to assess the effectiveness of a structured intervention on the frequency of self-care behaviors with AVF by patients with ESRD on hemodialysis (HD).

DETAILED DESCRIPTION:
This was a quasi-experimental study in dialysis units, involving patients using AVF for HD. The dialysis units are located in the north of Portugal (two units) and in the Autonomous Region of the Azores (one unit). The study started after approval by the institution ethics committee.

Study Setting and Population The study was carried out in dialysis units the north of Portugal, identified as Control Group (CG), and on an island in the Autonomous Region of the Azores, identified as Intervention Group (IG).

Data Collection and Instrument All data were collected from January to June 2018. Information concerning the sample demographic characteristics (age, gender, education, employment, marital status) and clinical characteristics (ESRD etiology, dialysis vintage, previous AVFs, AVF duration, information on care with the AVF) was collected with a questionnaire designed by the authors.

Information concerning self-care behaviors with the AVF was collected from the Scale of Assessment of Self-Care Behaviors with Arteriovenous Fistula in Hemodialysis (ASBHD-AVF) (8). This scale has 16 items in two subscales: subscale 1 - Management of Signs and Symptoms (6 items) and subscale 2 - Prevention of Complications (10 items). Responses to each item are based on a 5-point Likert-type scale. Higher scores show patients' higher frequency of self-care with the AVF. The ASBHD-AVF scale has been applied to Portuguese patients with Cronbach's alpha of 0.797, 0.797 and 0.722 for the global scale and sub-scales 1 and 2, respectively.

Memory problems were assessed by the Six-Item Cognitive Impairment Test (6CIT), Portuguese version (9).

ELIGIBILITY:
Inclusion Criteria:

* participants should be 18 years or older;
* have an AVF duration on HD greater than 6 months
* have no memory problems
* be medically stable.

Exclusion Criteria:

* patients with double vascular access (central venous catheter and AVF) or grafts as vascular access
* hospitalized patients at the time of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
scale of assessment of self-care behaviors with arteriovenous fistula in hemodialysis (ASBHD-AVF) | Change from baseline self-care behaviors at 12 months
  self-care behaviors with arteriovenous

SECONDARY OUTCOMES:
scale of assessment of self-care behaviors with arteriovenous fistula in hemodialysis (ASBHD-AVF) | Change from baseline self-care behaviors at 12 months
  Self-care behaviors with Management of signs and symptoms
scale of assessment of self-care behaviors with arteriovenous fistula in hemodialysis (ASBHD-AVF) | Change from baseline self-care behaviors at 12 months
  Self-care behaviors with prevention of complications

CONTACTS AND LOCATIONS:
Locations (1):
- clemente Sousa, Porto, Portugal

REFERENCES:
- [Derived] Sousa CN, Paquete ARC, Teles P, Pinto CMCB, Dias VFF, Ribeiro OMPL, Manzini CSS, Nicole AG, Souza LH, Ozen N. Investigating the Effect of a Structured Intervention on the Development of Self-Care Behaviors With Arteriovenous Fistula in Hemodialysis Patients. Clin Nurs Res. 2021 Jul;30(6):866-874. doi: 10.1177/1054773820974834. Epub 2020 Dec 3. PMID 33269608